CLINICAL TRIAL: NCT00502333
Title: The Influence of Coping Strategies and Catastrophizing on Patients With Back and Neck Pain Treated Within the Spanish National Health Service
Brief Title: The Influence of Coping Strategies and Catastrophizing on Patients With Back and Neck Pain
Status: Completed | Type: Observational
Sponsor: Kovacs Foundation (Other)
Responsible Party: Principal Investigator, Francisco M. Kovacs, Director of Scientific Department, Kovacs Foundation, Kovacs Foundation
Other Study IDs: FK-R-20
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Back Pain; Neck Pain
Keywords: back pain; neck pain; prognosis; catastrophizing; coping strategies; disability; Prognosis for back and neck pain
MeSH Terms: conditions — Back Pain; Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the influence of coping strategies and catastrophizing thoughts on disability and the prognosis of back and neck pain in patients treated within the Spanish National Health Service. Patients will be given a visual analog scale (VAS) to rate intensity of pain, the Roland Morris Questionnaire (RMQ) or the Neck Disability Index (NDI) to rate the degree of disability, and the Coping Strategies Questionnaire (CSQ) to rate coping strategies and catastrophizing. Questionnaires will be given at baseline and three months later.

ELIGIBILITY:
Inclusion Criteria:

* Subjects treated for back or neck pain in the Spanish National Health Service.
* Able to read and write Spanish.
* Have signed the informed consent form.

Exclusion Criteria:

* Diagnosis or "red flags" for systemic diseases (e.g., cancer, infection).
* Pain due to fracture or direct trauma to the neck or back.
* Criteria for referral to surgery (e.g., neurogenic claudication due to spinal stenosis, cauda equina syndrome, serious nerve root compression for more than 6 weeks due to disc herniation).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated within the Spanish National Health Service for subacute or chronic neck or back pain
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2006-11; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Disability | Baseline and 3 months

SECONDARY OUTCOMES:
Pain | Baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Director — Kovacs Foundation, Palma de Mallorca, 07012, Spain; Mario Gestoso, MD, Principal Investigator — Kovacs Foundation,Palma de Mallorca, Spain
Locations (1):
- Kovacs Foundation, Palma de Mallorca, Balearic Islands, Spain